CLINICAL TRIAL: NCT06515938
Title: Comparative Immunogenicity of Hepatitis B Vaccine With Different Immunization Schedule in Primary Immune Adults Aged 25-55 in China
Brief Title: Study on New Strategies for Hepatitis B Virus Immunization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wu Jiang (Other Government)
Responsible Party: Sponsor-Investigator, Wu Jiang, Director, Centers for Disease Control and Prevention, China
Organization: Centers for Disease Control and Prevention, China (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012ZX10002001
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Vaccine Reaction

ARMS (4):
- 20μg Engerix-B with 0-1-6 intervals (Experimental): Received three intramuscular injections of the 20μg Engerix-B vaccine with 0, 1, 6 month intervals
  Interventions: Biological: 20μg Engerix-B hepatitis B vaccine
- 20μg Kangtai with 0-1-6 intervals (Experimental): Received three intramuscular injections of the 20μg Kangtai hepatitis B vaccine with 0, 1, 6 month intervals
  Interventions: Biological: 20μg Kangtai hepatitis B vaccine
- 60μg Kangtai with 0-2 intervals (Experimental): Received two intramuscular injections of the 60μg Kangtai hepatitis B vaccine with 0, 2 month intervals
  Interventions: Biological: 60μg Kangtai hepatitis B vaccine
- 20μg CHO with 0-1-6 intervals (Placebo Comparator): Received three intramuscular injections of the 20μg Huabei hepatitis B vaccine made by recombinant DNA techniques in CHO cell with 0, 1, 6 month intervals
  Interventions: Biological: 20μg CHO

INTERVENTIONS:
Biological: 20μg Engerix-B hepatitis B vaccine
  Arms: 20μg Engerix-B with 0-1-6 intervals
Biological: 20μg Kangtai hepatitis B vaccine
  Arms: 20μg Kangtai with 0-1-6 intervals
Biological: 60μg Kangtai hepatitis B vaccine
  Arms: 60μg Kangtai with 0-2 intervals
Biological: 20μg CHO
  Arms: 20μg CHO with 0-1-6 intervals

SUMMARY:
To investigate the immunogenicity of HB vaccine with different series among primary immune adults aged 25-55, to assess potential alternative approaches for HB immunization.

DETAILED DESCRIPTION:
By comparing the immunization effect of hepatitis B vaccine with other different types of hepatitis B vaccines using seris procedure, information on the immunization effect of 60 micrograms of hepatitis B vaccine in adults was obtained, which will provide a scientific basis for the development of a rapid immunization procedure for adults with large doses of hepatitis B vaccine and for the improvement of the immunization strategy for hepatitis B in adults.

ELIGIBILITY:
Inclusion Criteria:

* aged 25-55 years
* negative for HBsAg,anti-HBs, and anti-HBc without prior HBV or HAV vaccination

Exclusion Criteria:

* a history of vaccine component allergies
* autoimmune diseases
* immunodeficiency
* vaccinations received within the past month
* acute illnesses within the past week
* fever (axillary temperature exceeding 38°C) within the past three days

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1169 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Anti-HBs | at the second month after the final injection of each arm
  Titers of hepatitis B virus surface antibody

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, Principal Investigator — Beijing Center for Disease Control and Prevention
Locations (2):
- China (2):
  - Huaibei District Center for Disease Control and Prevention, Huaibei, Anhui
  - Xuanhua District Center for Disease Control and Prevention, Xuanhua, Hebei

IPD SHARING:
Plan to Share IPD: Yes
The original primary outcome data will be shared
Supporting Information: Study Protocol
Time Frame: the data will become available after publication permanent
Access Criteria: With consent of the principal investigator